CLINICAL TRIAL: NCT02923258
Title: Postoperative Radiation and Concurrent Chemotherapy With Weekly Docetaxel Versus Cisplatin in Patients With High-risk Oral Cavity Cancer: a Randomized Phase II Clinical Trial
Brief Title: Postoperative CCRT With Docetaxel vs Cisplatin in High Risk Oral Cavity Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, MD, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016HNRT004
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
Keywords: oral cavity squamous cell carcinoma; concurrent chemotherapy; High-Risk
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Concurrent Chemoradiotherapy With Docetaxel and IMRT
  Interventions: Drug: Docetaxel; Radiation: IMRT
- Control (Active Comparator): Concurrent Chemoradiotherapy With Cisplatinum and IMRT
  Interventions: Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: Docetaxel — 20mg/m2/w
  Arms: Experimental
Drug: Cisplatin — 100mg/m2/q3w
  Arms: Control
Radiation: IMRT — a total dose of 60Gy in 30fractions over 6 weeks

SUMMARY:
This is a randomized,controled, phase II, open label study of postoperative concurrent chemoradiotherapy with Docetaxel versus Cisplatin for high-risk squamous cell carcinoma of the oral cavity cancer.The primary purpose of this study is to evaluate the efficacy of concurrent chemoradiotherapy with docetaxel in OCC patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically confirmed squamous cell carcinoma of the oral cavity 2. Gross total resection, with pathology demonstrating one or more of the following risk factors:

  1. Histologic extracapsular nodal extension
  2. Histologic involvement of ≥ 2 regional lymph nodes
  3. Invasive cancer is seen on microscopic evaluation of the resection margin, with no evidence of gross tumor residual 3. No evidence of distant metastases 4. No synchronous or concurrent head and neck primary tumors 5. ECOG 0-1 6. Adequate organ function including the following:

  <!-- -->

  1. Absolute neutrophil count (ANC) >= 1.5 * 10^9/l
  2. Platelets count >= 100 * 10^9/l
  3. Hemoglobin >= 10 g/dl
  4. AST and ALT <= 2.5 times institutional upper limit of normal (ULN)
  5. Total bilirubin <= 1.5 times institutional ULN
  6. Creatinine clearance >= 50 ml/min
  7. Serum creatine <= 1 times ULN 7.Signed written informed consent

Exclusion Criteria:

* 1. Evidence of distant metastasis 2. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region 3. Other previous cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma 4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures 5.Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  the time in months between the date of random assignment and the date of death from any cause
Locoregional failure-free survival (LRFS) | 2 years
  the time in months between random assignment and the date of first locoregional recurrence or death from any cause, whichever occurred first
distant metastasis free survival (DMFS) | 2 years
  the time from random assignment to the first distant metastasis or death from any cause
Adverse Events (AE) | 3 months
  AEs were summarized and recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Zhu, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang W, Chen L, Li R, Li J, Dou S, Ye L, He Y, Tian Z, Yao Y, Zhu G. Postoperative radiotherapy with docetaxel versus cisplatin for high-risk oral squamous cell carcinoma: a randomized phase II trial with exploratory analysis of ITGB1 as a potential predictive biomarker. BMC Med. 2024 Jul 29;22(1):314. doi: 10.1186/s12916-024-03541-6. PMID 39075531